CLINICAL TRIAL: NCT03554174
Title: Psilocybin - Induced Neuroplasticity in the Treatment of Major Depressive Disorder
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Heffter Research Institute (Other)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2000022394
Record Dates: First submitted 2018-04-13; First posted 2018-06-13 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder
Keywords: psilocybin
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo/Low Dose Psilocybin (Experimental): Subjects in this arm receive placebo in the first session and low dose psilocybin in the second session.
  Interventions: Drug: Low Dose Psilocybin; Drug: Placebo
- Placebo/Medium Dose Psilocybin (Experimental): Subjects in this arm receive placebo in the first session and medium dose psilocybin in the second session.
  Interventions: Drug: Placebo; Drug: Medium Dose Psilocybin
- Low Dose Psilocybin/Placebo (Experimental): Subjects in this arm receive low dose psilocybin in the first session and placebo in the second session.
  Interventions: Drug: Low Dose Psilocybin; Drug: Placebo
- Medium Dose Psilocybin/Placebo (Experimental): Subjects in this arm receive medium dose psilocybin in the first session and placebo in the second session.
  Interventions: Drug: Placebo; Drug: Medium Dose Psilocybin

INTERVENTIONS:
Drug: Low Dose Psilocybin — 0.1 mg/kg psilocybin capsule
  Arms: Low Dose Psilocybin/Placebo; Placebo/Low Dose Psilocybin
Drug: Placebo — microcrystalline cellulose capsule
Drug: Medium Dose Psilocybin — 0.3 mg/kg psilocybin capsule
  Arms: Medium Dose Psilocybin/Placebo; Placebo/Medium Dose Psilocybin

SUMMARY:
The primary goal of this pilot study is to investigate whether psilocybin alters neuroplasticity in people with major depressive disorder. The primary hypothesis is that psilocybin will result in neuroplastic changes that parallel improvement in symptoms of depression.

DETAILED DESCRIPTION:
In this placebo-controlled, blinded study, individuals with depression will participate in 2 experimental sessions approximately 4 weeks apart during which they will receive two of the following three interventions: 1) placebo, 2) low dose psilocybin (0.1 mg/kg), and 3) medium dose psilocybin (0.3 mg/kg).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Major Depressive Disorder (MDD), single or recurrent episode, and currently experiencing a Major Depressive Episode (MDE)
* Failed to achieve a satisfactory clinical response to at least one adequate antidepressant trial during the current depressive episode
* Currently engaged in treatment with a mental health clinician

Exclusion Criteria:

* Axis I psychotic disorder (e.g. schizophrenia, bipolar I, depression with psychosis)
* Axis I psychotic disorder in first degree relative
* Currently taking a conventional antidepressant medication
* Unstable medical or neurological conditions
* Significant cognitive disorders
* History of intolerance to drugs known to significantly alter perception e.g., psilocybin, LSD, salvinorin A, mescaline, etc.
* Pregnant, breastfeeding, lack of adequate birth control
* Urine toxicology positive to drugs of abuse on experimental test days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Changes in electrical brain activity associated with neuroplasticity measured by Electroencephalography (EEG) | One day and two weeks after each experimental session
  An auditory Long Term Potentiation (LTP) task will assess changes in neuroplasticity. For the EEG task, the outcome measures will include stimulus-evoked time x frequency analysis (e.g., spectral power)

SECONDARY OUTCOMES:
Changes in verbal memory [ Time Frame: One day and two weeks after each experimental session ] | One day and two weeks after each experimental session
  This will be measured by a modified computer version of the Rey Auditory Verbal Learning Test (RAVLT), administered while EEG data is collected. The EEG outcomes will include time x frequency analysis (e.g., spectral power) during the learning and recognition phases of the task.
Change in mood symptoms using the GRID-Hamilton Depression Rating Scale (GRID-HAM-D) | Four weeks before the initiation of testing, the day before and after each experimental session, and one and two weeks after each experimental session.
  The GRID-Hamilton Depression Rating Scale is a clinician-administered rating scale designed to assess severity of depressive symptoms. It includes 17 items, nine of which are scored on 5-point scale, and eight of which are scored on a three-point scale. The score range for the GRID-HAMD is 0 to 52, with higher score indicating more severe depression.
Change in mood symptoms using the Quick Inventory of Depressive Symptoms (QIDS-SR16) | Four weeks before the initiation of testing, the day before and after each experimental session, one and two weeks after each experimental session, then monthly for three months after the last experimental session.
  The QIDS-SR16 is a 16-item self-reported rating scale designed to assess severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak D'Souza, MD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven Campus, West Haven, Connecticut, United States